CLINICAL TRIAL: NCT00208793
Title: Calcium, Vitamin D, and Colon Cancer Risk Biomarkers
Brief Title: Calcium and Vitamin D vs Markers of Adenomatous Polyps
Acronym: CaDvMAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Roberd Bostick, MD, MPH, Professor, Emory University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0126-2004; R01CA104637 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Colorectal Adenomatous Polyps
Keywords: colonic polyps; adenomatous polyps; colon cancer prevention; dietary supplements
MeSH Terms: conditions — Colonic Polyps; Adenomatous Polyps | interventions — Calcium; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Calcium (Experimental): Calcium 2,000 mg/day as calcium carbonate in two divided doses with food
  Interventions: Dietary Supplement: Calcium
- Vitamin D3 (Experimental): Vitamin D3 800 IU given as 400 IU twice daily with food over 6 months
  Interventions: Dietary Supplement: Vitamin D3
- Calcium and vitamin D3 combined (Experimental): Calcium 2,000 mg (as calcium carbonate) + vitamin D3 800 IU given in equal divided doses twice daily with meals over 6 months
  Interventions: Dietary Supplement: Calcium and vitamin D3 combined
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Calcium and vitamin D3 combined — Calcium 2,000 mg (as calcium carbonate) + vitamin D3 800 IU given in equal divided doses twice daily with food over 6 months
  Arms: Calcium and vitamin D3 combined
Drug: Placebo — Placebo
  Arms: Placebo
Dietary Supplement: Calcium — Calcium 2,000 mg/day as calcium carbonate in two divided doses with meals over 6 months
  Arms: Calcium
Dietary Supplement: Vitamin D3 — Vitamin D3 800 IU given as 400 IU twice daily with food over 6 months
  Arms: Vitamin D3

SUMMARY:
The purpose of this study is to test whether calcium and/or vitamin D supplementation favorably affects a set of biomarkers of risk for colon cancer in persons who are at higher than average risk for colon cancer (ie, have already undergone the removal of adenomatous polyps, which are known to be precursors to developing colon cancer).

DETAILED DESCRIPTION:
There is strong biologic plausibility and animal experimental evidence for protection against colorectal cancer by calcium and vitamin D, calcium significantly reduced adenoma recurrence in a large clinical trial in humans (yet the previously reported observational evidence, although generally supportive, is inconsistent), and the observational literature strongly supports protection from vitamin D. A close physiological relationship between calcium and vitamin D has long been known. Yet, other than a possible reduction of colorectal epithelial cell proliferation by calcium, the effects of calcium and vitamin D, individually or jointly, on the normal human colorectal epithelium remain unknown. There have been no clinical trials involving vitamin D individually or jointly with calcium related to colorectal cancer chemoprevention in humans. There are currently no generally accepted pre-neoplastic biomarkers of risk for colorectal cancer other than the possible exception of proliferation markers that, at best, have limited usefulness as individual markers. Based on recent advances in understanding the molecular basis of colorectal cancer, we developed a panel of newer, plausible, reliable, immunohistochemically detected biomarkers that provides molecular phenotyping of the normal appearing colorectal epithelium: 1) inflammation (COX-2), 2) the expression of genes involved in the normal structure and function of the colorectal epithelium that have been found to be altered early in the two major colorectal carcinogenesis pathways (APC, MSH2, MLH1), and 3) a more complete picture of the cell cycle events in colorectal epithelial crypt cells (short and long-term proliferation: MIB-1 and telomerase; differentiation: p21; apoptosis inhibition and promotion: bcl-2, bax, and bak) that has not yet been tested in a chemoprevention trial.

To address these needs, we will conduct a preliminary, randomized, double-blind, placebo-controlled, 2 x 2 factorial chemoprevention trial (n = 88) of calcium 2,000 mg/day and vitamin D3 800 IU/day, alone and in combination vs placebo over 6 months in patients with recent removal of sporadic adenomatous colorectal polyps, to investigate their effects on the individual components and aggregate profile of our colorectal cancer risk biomarker panel. We will also examine study results stratified by NSAID use and Bsm I vitamin D receptor genotypes. The preliminary estimates of treatment effect sizes and variabilities will be used to refine the biomarker panel and study design and to calculate the needed sample size for a potential full-scale study.

We assert that using biological measurements of risk, as they have for ischemic heart disease, will result in a decline in colorectal cancer incidence and mortality. The proposed project is borne of this vision, and has intertwined missions of exploring the efficacy of two plausible and evidentially well-supported dietary agents, calcium and vitamin D, on the modulation of a plausible panel of molecular phenotypic biomarkers of risk for colorectal neoplasia.

ELIGIBILITY:
Inclusion Criteria:

* age 30-74
* adenomatous colon polyp within past 3 years
* general good health with life expectancy of at least 2 years
* available for 8 months and able to come for clinic visits

Exclusion Criteria:

* cancer within 5 years
* active major disease
* renal impairment
* history of kidney stones
* significant dietary change or weight loss within past 6 months
* unable to forego usual calcium or vitamin D use during study

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2005-05; Primary Completion 2006-09 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Biomarkers of Risk for Colorectal Neoplasms | 6 months
  A panel of putative biomarkers of risk for colorectal neoplasms in biopsies of normal appearing rectal mucosa: COX-2, APC, MSH-2, MLH1, MIB-1, telomerase, p21, bcl-2, bax, bak, β-catenin, E-cadherin, TGFα, TGFβ1, calcium sensing receptor, vitamin D receptor, CYP27B1, CYP24, 8-OH-dG

SECONDARY OUTCOMES:
Vitamin D metabolites | 6 months
  serum 25-OH-vitamin D3 and 1,25-OH-vitamin D3
Circulating inflammation markers | 6 months
  serum CRP, TNF-α, IL-6, IL-1β, IL-8 and IL-10

CONTACTS AND LOCATIONS:
Overall Officials: Roberd M Bostick, MD, MPH, Principal Investigator — Emory University, Rollins School of Public Health & Winship Cancer Institute
Locations (1):
- The Emory Clinic, Division of Digestive Diseases, Atlanta, Georgia, United States

REFERENCES:
- [Result] Fedirko V, Bostick RM, Flanders WD, Long Q, Shaukat A, Rutherford RE, Daniel CR, Cohen V, Dash C. Effects of vitamin D and calcium supplementation on markers of apoptosis in normal colon mucosa: a randomized, double-blind, placebo-controlled clinical trial. Cancer Prev Res (Phila). 2009 Mar;2(3):213-23. doi: 10.1158/1940-6207.CAPR-08-0157. Epub 2009 Mar 3. PMID 19258546
- [Result] Fedirko V, Bostick RM, Flanders WD, Long Q, Sidelnikov E, Shaukat A, Daniel CR, Rutherford RE, Woodard JJ. Effects of vitamin d and calcium on proliferation and differentiation in normal colon mucosa: a randomized clinical trial. Cancer Epidemiol Biomarkers Prev. 2009 Nov;18(11):2933-41. doi: 10.1158/1055-9965.EPI-09-0239. Epub 2009 Oct 27. PMID 19861511
- [Result] McCullough ML, Bostick RM, Daniel CR, Flanders WD, Shaukat A, Davison J, Rangaswamy U, Hollis BW. Vitamin D status and impact of vitamin D3 and/or calcium supplementation in a randomized pilot study in the Southeastern United States. J Am Coll Nutr. 2009 Dec;28(6):678-86. doi: 10.1080/07315724.2009.10719801. PMID 20516268
- [Result] Fedirko V, Bostick RM, Long Q, Flanders WD, McCullough ML, Sidelnikov E, Daniel CR, Rutherford RE, Shaukat A. Effects of supplemental vitamin D and calcium on oxidative DNA damage marker in normal colorectal mucosa: a randomized clinical trial. Cancer Epidemiol Biomarkers Prev. 2010 Jan;19(1):280-91. doi: 10.1158/1055-9965.EPI-09-0448. PMID 20056649
- [Result] Sidelnikov E, Bostick RM, Flanders WD, Long Q, Fedirko V, Shaukat A, Daniel CR, Rutherford RE. Effects of calcium and vitamin D on MLH1 and MSH2 expression in rectal mucosa of sporadic colorectal adenoma patients. Cancer Epidemiol Biomarkers Prev. 2010 Apr;19(4):1022-32. doi: 10.1158/1055-9965.EPI-09-0526. Epub 2010 Mar 23. PMID 20332274
- [Result] Ahearn TU, McCullough ML, Flanders WD, Long Q, Sidelnikov E, Fedirko V, Daniel CR, Rutherford RE, Shaukat A, Bostick RM. A randomized clinical trial of the effects of supplemental calcium and vitamin D3 on markers of their metabolism in normal mucosa of colorectal adenoma patients. Cancer Res. 2011 Jan 15;71(2):413-23. doi: 10.1158/0008-5472.CAN-10-1560. Epub 2010 Nov 17. PMID 21084270
- [Result] Hopkins MH, Owen J, Ahearn T, Fedirko V, Flanders WD, Jones DP, Bostick RM. Effects of supplemental vitamin D and calcium on biomarkers of inflammation in colorectal adenoma patients: a randomized, controlled clinical trial. Cancer Prev Res (Phila). 2011 Oct;4(10):1645-54. doi: 10.1158/1940-6207.CAPR-11-0105. Epub 2011 Jun 30. PMID 21724580
- [Result] Chai W, Bostick RM, Ahearn TU, Franke AA, Custer LJ, Cooney RV. Effects of vitamin D3 and calcium supplementation on serum levels of tocopherols, retinol, and specific vitamin D metabolites. Nutr Cancer. 2012;64(1):57-64. doi: 10.1080/01635581.2012.630552. Epub 2011 Dec 9. PMID 22149065
- [Result] Ahearn TU, Shaukat A, Flanders WD, Rutherford RE, Bostick RM. A randomized clinical trial of the effects of supplemental calcium and vitamin D3 on the APC/beta-catenin pathway in the normal mucosa of colorectal adenoma patients. Cancer Prev Res (Phila). 2012 Oct;5(10):1247-56. doi: 10.1158/1940-6207.CAPR-12-0292. Epub 2012 Sep 10. PMID 22964475
- [Result] Hopkins MH, Flanders WD, Bostick RM. Associations of circulating inflammatory biomarkers with risk factors for colorectal cancer in colorectal adenoma patients. Biomark Insights. 2012;7:143-50. doi: 10.4137/BMI.S10092. Epub 2012 Nov 5. PMID 23170065
- [Derived] Tu H, Flanders WD, Ahearn TU, Daniel CR, Gonzalez-Feliciano AG, Long Q, Rutherford RE, Bostick RM. Effects of calcium and vitamin D3 on transforming growth factors in rectal mucosa of sporadic colorectal adenoma patients: a randomized controlled trial. Mol Carcinog. 2015 Apr;54(4):270-80. doi: 10.1002/mc.22096. Epub 2013 Oct 26. PMID 24166893